CLINICAL TRIAL: NCT05073393
Title: Effect of Probiotics on Oral Homeostasis During Sugar Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: Deerland Probiotics and Enzymes (Unknown)
Responsible Party: Principal Investigator, Daniel Belstrøm, DDS, PhD, DDS, PhD, Dr. odont, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UCPH_01_005
Record Dates: First submitted 2021-10-08; First posted 2021-10-11 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Dental Caries; Probiotics; Gingivitis
MeSH Terms: conditions — Dental Caries; Gingivitis

STUDY DESIGN:
Intervention Model Description: Double blinded randomized clinical trial with a test and placebo group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Computerized randomization only known to the principal investigator, who are not directly involved in data collection or data analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): In this group participants will receive probiotic supplements twice a day (morning and evening) for at period of 28 days (14 days with sugar stress followed by 14 days without sugar stress).
  Interventions: Behavioral: Sugar stress
- Placebo (Placebo Comparator): In this group participants will receive placebo twice a day (morning and evening) for at period of 28 days (14 days with sugar stress followed by 14 days without sugar stress).
  Interventions: Behavioral: Sugar stress

INTERVENTIONS:
Behavioral: Sugar stress — Sucrose rinsing for 14 days (8-10 times a day) followed by 14 days without sucrose rinsing

SUMMARY:
The present study is a double-blinded randomized clinical trial with a duration of 28 days.

DETAILED DESCRIPTION:
The present study is a double-blinded randomized clinical trial with a duration of 28 days.

80 orally and systemically healthy participant will be allocated in the test (probiotic) and the control (placebo) group at baseline.

The intervention is sugar stress, which will be applied at baseline and continue through day 14, followed by 14 days without sugar stress.

Clinical measurements and sampling will be performed at baseline, day 14 and day 28

Primary endpoint: Changes in microbial composition.

Secondary endpoints: Changes in clinical and immunological parameters

ELIGIBILITY:
Inclusion Criteria:

* age > 18 yrs.

Exclusion Criteria:

* Presence of oral diseases i.e. gingivitis, periodontitis and dental caries
* Current smokers
* Any systemic diseases and current use of any medication with known effect on oral health
* Use of systemic antibiotics within the latest three months.
* Age < 18 yrs., and age > 30 yrs.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Changes in microbial composition in dental plaque | Baseline vs. Day 14 and Day 28
  Changes in alpha and beta diversity of microbial composition

SECONDARY OUTCOMES:
Changes in clinical parameters | Baseline vs. Day 14 and Day 28
  Changes in levels of dental plaque and gingival inflammation
Changes in salivary levels of inflammatory cytokines | Baseline vs. Day 14 and Day 28
  Changes in mean salivary levels of selected inflammatory cytokines

CONTACTS AND LOCATIONS:
Locations (1):
- University of Copenhagen, Department of Odontology, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No